CLINICAL TRIAL: NCT02480491
Title: Study of Cell Free DNA Content of Human Embryo Culture Medium as a Non-Invasive Tool for Embryo Assessment in ICSI Treatment Cycles
Brief Title: Study of Free DNA Content of Embryo Culture Medium as a Non-Invasive Tool for Embryo Assessment
Status: Completed | Type: Observational
Sponsor: Sadat City University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Azza Awad Abdel Razik Mohamed, Director of Embryology Lab., Ain Shams Univesity, Sadat City University
Other Study IDs: SCS-1
Record Dates: First submitted 2015-06-20; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — cell free DNA content of the culture medium of the human embryo
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Third day embryos: embryos culture media during third day after fertilization
  Interventions: Other: measuring cell freeDNA
- Fifth day embryos: embryos culture media during fifth day after fertilization
  Interventions: Other: measuring cell freeDNA

INTERVENTIONS:
Other: measuring cell freeDNA — measuring cell free DNA using PCR

SUMMARY:
Study of Cell Free DNA Content of Human Embryo Culture Medium as a Non-Invasive Tool for Embryo Assessment in intra cytoplasmic sperm injection Treatment Cycles.

DETAILED DESCRIPTION:
The aim of the present study is to determine whether cell free DNA content of the culture medium of the human embryo correlates with the quality and reproductive potential of embryos in ICSI cycles and, thus, to look for a new non invasive tool of assessing embryo quality beside morphological assessment. Determining a rapid, noninvasive method for the assessment of the developmental potential of embryos may be a great achievement

ELIGIBILITY:
Inclusion Criteria:

* third day embryos

Exclusion Criteria:

* less than third day embryos

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ICSI Treatment Cycles females
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
correlations between levels of measured cell free DNA and embryo quality. | 12 months